CLINICAL TRIAL: NCT04360499
Title: The Effect of a Three Month, Low- Load- High- Repetitions Group-based Exercise Program Versus Pilates on Physical Fitness and Body Composition in Inactive Women
Brief Title: Low- Load- High- Repetitions Training Versus Pilates on Physical Fitness in Inactive Women
Acronym: GetActive
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Thessaly (Other)
Collaborators: University of Nicosia (Other)
Responsible Party: Principal Investigator, Giorgos K. Sakkas, Professor, University of Thessaly
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: EEBK/EΠ/2015/34
Record Dates: First submitted 2020-04-13; First posted 2020-04-24 (Actual); Last update posted 2021-10-06 (Actual); Status verified 2021-09

CONDITIONS: Sedentary Behavior
Keywords: fitness; body fat; trunk fat; sleep; Pilates; Women
MeSH Terms: conditions — Sedentary Behavior | interventions — Exercise Movement Techniques

STUDY DESIGN:
Intervention Model Description: Participants will be randomly allocated in two groups: the LLHR group and the Pilates group. Both exercise programs will be performed in groups lasting for three months and performed 3 times per week.
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants will not be aware of the type of exercise intervention. Assessors will be blind for the group allocation of the participants
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low-weight-high-repetitions training (Experimental): Low-weight-high-repetitions (LWHR) refer to a specific form of resistance exercise which utilizes low weights and very high repetitions. Participants will be exercised 3 times per week for 3 months in small groups.
  Interventions: Other: Low- weight-high-repetitions training
- Pilates Training (Active Comparator): Pilates exercises focused on breathing, concentration, control and precision. Participants will be exercised 3 times per week for 3 months in small groups
  Interventions: Other: Pilates training

INTERVENTIONS:
Other: Low- weight-high-repetitions training — LWHR refers to a specific form of resistance exercise which utilizes low weights and very high repetitions
  Arms: Low-weight-high-repetitions training
Other: Pilates training — Pilates style exercise training
  Arms: Pilates Training

SUMMARY:
Low-weight-high-repetitions (LWHR) programs constitute a popular group-based form of exercise for the general population, accompanied by various health benefits for the participants. However, the effect of such programs on cardiorespiratory fitness is still controversial. The aim of the current study was to examine the effects of a 3-month LWHR group exercise program vs pilates on cardiorespiratory fitness, body composition and overall health on previously inactive adult women.

DETAILED DESCRIPTION:
This is a randomized exercise intervention study in healthy subjects (adult women-inactive). Participants will be randomly allocated in two groups: the LLHR group and the Pilates group. All assessments will be blinded to the intervention group of the participants. Both exercise programs will be performed in groups lasting for three months and performed 3 times per week. The study conformed to the principles enumerated in the Helsinki Declaration and ethical approval has been obtained by the national ethical committee.

Participants in the LLHR training will participate in a three-month, group based pre-choreographed exercise programme, consisting of three LLHR training sessions per week (in non-consecutive days). All participants will be familiar with the exercises that will be used in this intervention. Each LLHR fitness program, includes a variety of multifunction exercises (i.e. squats, lunges, chest press and chest extension, rowing, triceps extension and bicep curls) addressing all muscle groups; using barbells, dumbbells or body weight. Each session will last for 60 min (including 5 min warm up and 5 min cooldown). Exercise intensity will increase progressively once a month by adding weights to the barbells and dumbbells.

Participants in the Pilates program will be trained with the same exercise schedule for the 3-month period. Their 60 min session, will be consisted of warm-up and cool down (5 minutes each), along with static-isometric exercises addressing major muscle groups. Pilates exercises focus on breathing, concentration, control and precision. Exercise intensity progression in the Pilates program will be performed every one month by increasing the level of demanding of the exercises.

All training sessions of both the LLHR and Pilates programs will be supervised by a qualified sports scientist (one sport scientist responsible for each program) for securing training standardization. Participants in both programs will be advised to avoid taking part in any other exercise session during the intervention period.

ELIGIBILITY:
Prior to the initiation of the study, participants will be examined by a physician for confirming their health status. According to the updated criteria, "inactive" is an individual who is performing insufficient amounts of moderate-to-vigorous physical activity (Sedentary Behaviour Research Network, 2012).

Inclusion Criteria:

* Female, inactive, able to participate in an exercise training

Exclusion Criteria:

* male gender, inability to perform the exercise training program due to musculoskeletal injury, a medication that could affect cardio-metabolic function, including anti-hypertensive, diabetic or anti-obesity drugs and inability to systematically participate in the proposed training programs according to the schedule (i.e. absence from 3 consecutive exercise sessions or missed more than 10% of total exercise sessions), psychiatric disorders.

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Inactive but otherwise healthy adult women will participate in the current study.
Enrollment: 60 (Actual)
Dates: Start 2018-01-10 (Actual); Primary Completion 2020-08-10 (Actual); Study Completion 2021-09-10 (Actual)

PRIMARY OUTCOMES:
Changes from baseline Aerobic Fitness at 12 weeks | 12 weeks
  The 20m shuttle run will be used in order to assess aerobic fitness levels (Leger et al., 1988). Briefly, the 20m shuttle run test involves continuous shuttle running, between two parallel lines set exactly at 20m apart, in time to recorded beeps being indicated by signals produced from a commercially available pre-recorded CD (Coachwise Ltd, UK). Initial speed dictated at 8.5 km/h and increased by 0.5 km/h per minute. The test for each participant will be terminated when the participant could no longer maintain the speed-pace, for more than two consecutive beeps. For each participant, the number of shuttles completed will be recorded as an index of their aerobic fitness level (Leger et al., 1988).

SECONDARY OUTCOMES:
Changes from baseline Body Composition at 12 weeks | 12 weeks
  Body fat percentage will be measured using bioelectrical impedance analysis (BIA) (Tanita body composition analyser, TBF-300). Participants will be asked to avoid any fitness activity, caffeine consumption or eating for 3 hours previous to the test.

OTHER OUTCOMES:
Changes from baseline Muscle Strength at 12 weeks | 12 weeks
  Handgrip strength (in kg) of both arms will be measured using a digital dynamometer (T.K.K. 5401 Grip-D; Takey, Tokyo, Japan). For each arm, the participants will be asked to hold squeeze it for about 3 seconds, whilst no other movement was allowed.

CONTACTS AND LOCATIONS:
Overall Officials: Chistoforos Giannaki, PhD, Principal Investigator — University of Nicosia
Locations (1):
- U-Fit, Nicosia, Cyprus

IPD SHARING:
Plan to Share IPD: No
Only with other researchers participating in the study

REFERENCES:
- [Background] Evangelou C, Sakkas GK, Hadjicharalambous M, Aphamis G, Petrou P, Giannaki CD. The effect of a three month, low-load- high-repetitions group-based exercise program versus pilates on physical fitness and body composition in inactive women. J Bodyw Mov Ther. 2021 Apr;26:18-23. doi: 10.1016/j.jbmt.2020.08.017. Epub 2020 Sep 4. PMID 33992241